CLINICAL TRIAL: NCT04820634
Title: Using Virtual Reality to Improve Job Reentry in Adults With TBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-1090-19
Record Dates: First submitted 2021-02-03; First posted 2021-03-29 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-JIT (Experimental): In this arm, participants would participate in simulated interviews utilizing a software program and virtual interviewer, once a week for 90 minutes.
  Interventions: Other: Virtual Reality Job Interview Training
- Wonderworks (Placebo Comparator): In this arm, participants would participate in a similar intervention, also once a week for 90 minutes. However, in this arm, the intervention would be in a virtual office environment completing office tasks.
  Interventions: Other: Wonderworks

INTERVENTIONS:
Other: Virtual Reality Job Interview Training — The treatment group (TX) will complete 7 sessions of VR-JIT (1 sessions per week for 7 weeks), designed to teach the skills & concepts of job interviews. Sessions are approximately 90 minutes long.
  Arms: VR-JIT
Other: Wonderworks — The control group (CT) will complete 7 sessions of Wonderworks (1 session per week for 7 weeks) using skills in an office environment.
  Arms: Wonderworks

SUMMARY:
The purpose of this research is to investigate the effectiveness of virtual reality (VR) to improve job reentry skills in individuals with TBI.

DETAILED DESCRIPTION:
The current study will examine a virtual reality (VR) intervention entitled "Virtual Reality Job Interview Training (VR-JIT)" which targets social competency skills needed for successful job interviewing, and its efficacy when applied to individuals with traumatic brain injury (TBI). Preliminary evidence suggests that the VR-JIT is successful in individuals with autism spectrum disorder and schizophrenia in improving interview abilities. However, the efficacy of VR-JIT has not been evaluated in TBI populations.

ELIGIBILITY:
Inclusion Criteria:

* I am between the ages of 18 and 65.
* I have a diagnosis with moderate to severe TBI.
* I am at least one year post injury.
* I am able to speak and read English fluently.

Exclusion Criteria:

* I have a history of multiple sclerosis, stroke, seizures or another neurological injury or disease in the past (like brain tumor or epilepsy).
* I have a history of significant psychiatric illness (like bipolar disorder, schizophrenia or psychosis).
* I am currently taking steroids and/or benzodiazepines as determined by study staff review of my medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2024-07-28 (Estimated); Study Completion 2024-07-28 (Estimated)

PRIMARY OUTCOMES:
Change in Mock Job Interview Score at 1 month | 1 month
  Participants will complete a mock job interview at follow-up which will be compared to their initial interview and rated by blinded assessors on their job interview performance.

CONTACTS AND LOCATIONS:
Overall Officials: John DeLuca, Ph.D., Study Chair — Lab Director
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No